CLINICAL TRIAL: NCT01418196
Title: Relation of Diet to Heart Disease Risk Factors in Children
Status: Completed | Type: Observational
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Other Study IDs: MM-3462
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Healthy; Cardiovascular Disease
Keywords: TMAO; Children; Dietary choline; Cardiovascular disease risk; Atherogenic dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Metabolites of dietary phosphatidylcholine- choline and trimethylamine N-oxide (TMAO)- were recently identified as being associated with myocardial infarction in a case-control study. The latter TMAO is a gut-microflora-derived choline metabolite that has been shown to be a potent risk factor for cardiovascular disease (CVD). This pilot study seeks to use information derived from a dietary questionnaire in children to test the association of dietary choline intake to plasma levels of TMAO as well as the relationship between plasma choline levels and components of atherogenic dyslipidemia (increased triglycerides and small LDL, and reduced HDL cholesterol). An ancillary goal of this study is to build on existing programs of community outreach to local Oakland/Berkeley minority communities, and to develop an infrastructure for family-based and community participation in clinical research across the full age spectrum and among diverse populations. This pilot study will examine the association of dietary choline intake assessed by food frequency questionnaires to biomarkers of CVD risk in 40 children (> 7 years of age) and their parents as there is no information regarding this relationship in children. The results of this pilot study will form the basis for a proposal to carry out a randomized intervention trial to directly test the effects of dietary choline intake on plasma TMAO and lipoprotein levels. Ultimately, better understanding of the relationship between dietary choline intake and CVD risk factors may facilitate the formulation of appropriate dietary choline recommendations in children and adults.

DETAILED DESCRIPTION:
From interested participants (children and parents) we will obtain:

1. Informed consent
2. Anthropometric measurements - height, weight, waist and hip circumference, blood pressure, % body fat by bioimpedance (Tanita scale).
3. Health History Questionnaire
4. Food Frequency Questionnaire
5. Fasting blood sample- We will collect a total of 40 ml of blood (less than 3 ml/kg for the entire study). The blood samples will be used to measure triglyceride, LDL-cholesterol, HDL-cholesterol, glucose, insulin, apoA1, apoB, C-reactive protein, lipoprotein subfraction analysis by ion mobility, DNA for inclusion in our DNA biobank, choline, TMAO and other metabolites related to heart disease risk.

Standard Blood sampling: Using standard blood collection procedures, blood samples will be collected from participants after a 12-14 hour fast. The blood will be collected in tubes containing the following preservative solution: 3.0 gms EDTA (dipotassium), 1.7 mg P-Pack, 0.15 gms gentamycin sulfate, 0.15 gms chloramphenicol, 5.96 mls aprotinin (Sigma A-6279), and 0.30 gms sodium azide all of which are diluted to 20mls with doubly deionized water. Plasma is separated by immediate centrifugation at 4°C. Lipid and lipoprotein measurements are performed and aliquots of plasma are frozen for future analyses.

ELIGIBILITY:
Inclusion Criteria:

* Children >7 years of age and their parents

Exclusion Criteria:

* Antibiotics
* Pregnant or breastfeeding women

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of children (>7 years of age) and their parents who are generally healthy. Parents are not required to participant in the study. We will include all ethnicities.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Trimethylamine N-oxide (TMAO) | 1 time

SECONDARY OUTCOMES:
Choline | 1 time
LDL subfractions | 1 time
HDL cholesterol | 1 time
Triglycerides | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States